CLINICAL TRIAL: NCT05171595
Title: Real Time ST-segment Deviation Detection in High-risk Patients Detected by Wireless Single-lead ECG
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jonathan Attilla Koefoed Starling, Medical Student, Rigshospitalet, Denmark
Other Study IDs: ST-Deviation WARD
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Injury
Keywords: ST-deviations; Continuous wireless monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- no myocardial injury: In this study, patients were divided into groups of myocardial injury, where patients had TnT elevations (of 20-64 ng/L with an absolute change of ≥ 5 ng/L, or a hsTnT level ≥65 ng/L, both evaluated as due to ischemic etiology) and a group with no myocardial injury.
  Interventions: Device: Lifetouch single-lead ECG monitoring; Diagnostic Test: high-sensitive TnT measurements
- Myocardial injury: In this study, patients were divided into groups of myocardial injury, where patients had TnT elevations (of 20-64 ng/L with an absolute change of ≥ 5 ng/L, or a hsTnT level ≥65 ng/L, both evaluated as due to ischemic etiology) and a group with no myocardial injury.
  Interventions: Device: Lifetouch single-lead ECG monitoring; Diagnostic Test: high-sensitive TnT measurements

INTERVENTIONS:
Device: Lifetouch single-lead ECG monitoring — The continuous wireless monitoring is a single-lead ECG patch (Isansys Life Touch patch) which consists of two ECG electrodes placed on the left side of the patients' thorax. The patch measures respiratory rate (RR), heart rate (HR), heart rate variability (HRV) and electrocardiogram (ECG)s.
Diagnostic Test: high-sensitive TnT measurements — Another monitoring device in the study was the plasma concentration of high-sensitive cardiac troponin T (hsTnT).

SUMMARY:
This study primarily aims to describe the frequency of significant ST-deviations, defined as ECG-ST-deviations <-0.255 or >0.245 mV for a minimum duration of 30 minutes as measured by a single-lead ECG in patients admitted with AECOPD or following major abdominal surgery. Secondarily we will describe the frequency of ST-deviations <-0.255 or >0.245 mV for a minimum duration of 1, 10 and 20 minutes, respectively, as well as for patients with ST-deviations <-0.1 or >0.1 mV for a minimum duration of 1, 10, 20 and 30 minutes, respectively. Lastly, we will investigate the association between ST-deviations and subsequent myocardial injury while adjusting for known risk factors.

DETAILED DESCRIPTION:
Background:

Assesment of wireless ECG-monitoring devices is essential for patient monitoring as it enables activity and out-of-hospital monitoring. Former studies have found a random variation for ST-deviations between wireless single-lead ECG and 12-lead ECG, which suggests that clinical monitoring of ST-deviations by single-lead ECG must be corrected for this to minimize false positive cases. Thus, we aimed to assess how a corrected limit of agreement for ST-deviations affects the ability to detect true myocardial ischemia by comparing thresholds to troponin elevations.

Methods:

This study sought to analyze data from two WARD cohort studies (NCT03491137) and (NCT03660501). Patients were included at Rigshospitalet and Bispebjerg Hospital from February 2018 to September 2020. The Surgery and COPD studies consisted of 505 and 202 patients, respectively, who were hospitalized with AECOPD or scheduled for elective major abdominal surgery lasting > 2 hours. All patients were monitored with wireless equipment, which continuously measured vital signs. The continuous wireless monitoring used in this study consisted of a single-lead ECG patch (Isansys Life Touch patch) which consists of two ECG electrodes placed on the left side of the patients' thorax. The patch measures respiratory rate (RR), heart rate (HR), heart rate variability (HRV) and electrocardiogram (ECG)s. Another monitoring device was the plasma concentration of high-sensitive cardiac troponin T (hsTnT, Cobas 8000, e801 module, Diagnostics Roche). In this study, patients were divided into a myocardial injury group with TnT elevations (of 20-64 ng/L with an absolute change of ≥ 5 ng/L, or a hsTnT level ≥65 ng/L, both evaluated as due to ischemic etiology) and a group with no myocardial injury.

Analysis:

Baseline characteristics of patients undergoing major abdominal surgery and patients admitted with AECOPD with and without myocardial injury will be summarized in frequency tables including Using descriptive statistics, we will describe the occurrence of ST-segment deviations in the single-lead (Lifetouch) ECG in patients with and without myocardial injury as well as the association between ST-deviation and subsequent myocardial injury, which will be adjusted for known risk factors; age, gender, BMI, daily smoker (never-, previous-, current smoker), alcohol consumption (none, below- or above recommendations), ASA classification (ASA 1,2,3,4), history of myocardial infarction, history of diabetes mellitus, history of chronic heart failure. Furthermore, the sensitivity and specificity of continuous wireless single-lead ECG with the applied threshold of <-0.255 mV and > 0.245 mV will be determined. Receiver operating characteristics (ROC) analyses will be made to determine which type of ST-deviation and which specific threshold value was most sensitive for TnT elevations. Through ROC analyses it will also be examined how different variations of durations affect the thresholds' sensitivity and specificity. Statistical analysis will be performed using statistical software SPSS.

ELIGIBILITY:
Inclusion Criteria:

WARD-COPD:

* ≥ 18 years
* Patients admitted to emergency departments or pulmonary wards with AECOPD as admission diagnosis with suspected acute exacerbation of COPD
* The diagnosis had to be sustained in the patient record at the time of inclusion
* Expected admittance longer than 24 hours
* Possibility of an investigator to include the patient within 24 hours from admission

WARD-Surgery:

* ≥ 60 years
* Elective major abdominal cancer surgery
* Estimated surgical duration ≥ 2 hours.

Exclusion Criteria:

WARD-COPD:

* Patients who were not expected to cooperate to wear the monitoring equipment
* Unable to give informed consent
* Patients who were withheld active treatment
* Implanted cardioverter defibrillator or pacemaker
* Severe allergy for plaster/silicone

WARD-Surgery:

* Implanted cardioverter defibrillator or pacemaker
* Allergy to study devices
* Severe cognitive impairment assessed by MMSE
* Inability to cooperate wearing the wireless monitoring equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the two WARD studies: WARD COPD and WARD Surgery. Patients were included at Rigshospitalet (department of abdominal surgery) and Bispebjerg Hospital (departments of emergency medicine, pulmonary medicine, and abdominal surgery) in Denmark from February 2018 to September 2020 after obtained written informed consent. Eligibility was determined by the investigator. All patients were monitored with wireless equipment, which continuously measures vital signs.
Sampling Method: Non-Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with ST-deviation <-0.255 and/or >0.245 mV on single-lead ECG | 30 minutes
  The primary outcome is the frequency of patients with ST-deviation <-0.255 and/or >0.245 mV (0.1 mV + LoA) on single-lead ECG monitoring lasting ≥ 30 minutes.

SECONDARY OUTCOMES:
Frequency of patients with significant ST-deviations <-0.1 and/or >0.1 mV lasting ≥ 1 minute. | 1 minute
Frequency of patients with significant ST-deviations <-0.1 and/or >0.1 mV lasting ≥ 10 minutes. | 10 minutes
Frequency of patients with significant ST-deviations <-0.1 and/or >0.1 mV lasting ≥ 20 minutes. | 20 minutes
Frequency of patients with significant ST-deviations <-0.1 and/or >0.1 mV lasting ≥ 30 minutes. | 30 minutes
Frequency of patients with ST-deviation <-0.255 and/or >0.245 mV lasting ≥ 1 minute. | 1 minute
Frequency of patients with ST-deviation <-0.255 and/or >0.245 mV lasting ≥ 10 minutes. | 10 minutes
Frequency of patients with ST-deviation <-0.255 and/or >0.245 mV lasting ≥ 20 minutes. | 20 minutes
Frequency of patients with ST-deviation <-0.255 and/or >0.245 mV lasting ≥ 30 minutes and myocardial injury within three days of the first continuous monitoring day. | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Department of Anesthesiology, Centre for Cancer and Organ Diseases, University of Copenhagen, Blegdamsvej 9, 2200 Copenhagen, Denmark, Copenhagen, Denmark